CLINICAL TRIAL: NCT00325741
Title: Allogeneic Hematopoietic Cell Transplantation for Patients With Life-Threatening Systemic Lupus Erythematosus Using a Non-Myeloablative Regimen of Total Lymphoid Irradiation and Anti-Thymocyte Globulin
Brief Title: Allogeneic Blood Stem Cell Transplantation for Patients With Life-Threatening Systemic Lupus Erythematosus
Acronym: SLE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty with recruiting participants
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); City of Hope National Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 368; P01HL075462-02 (NIH)
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus; Systemic Lupus Erythematosus; Blood Stem Cell Transplantation
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietc Stem Cell Transplant (Experimental): Hematopoietic Cell Transplantation. Total body irradiation and Stem cell infusion in life threating lupus patients
  Interventions: Drug: Hematopoietic Cell Transplantation

INTERVENTIONS:
Drug: Hematopoietic Cell Transplantation — 1200 cGy total lymphoid irradiation (TLI) are administered on day -11 through -7 and days -4 through -1 pretransplantation; rabbit ATG at 1.5 mg/kg i.v. on days -11 through -7 pretransplantation; one single infusion of donor CD34+ cells plus selected T cell add back on completion of TLI (day 0); mycophenolate mofetil (MMF) is begun on day 0 at a dose of 15 mg/kg bid and stopped on day +28; cyclosporine (CSP) at initial dose of 6.25 mg/kg and adjusted to maintain trough blood levels of 350-500 ng/ml is begun on day -3 to complete withdrawal by 6 months post-transplantation.
  Other Names: NCT00325741

SUMMARY:
The Stanford Medical Center Division of Immunology and Rheumatology and the Division of Blood and Marrow Transplantation (BMT) are enrolling patients with severe systemic lupus erythematosus (SLE) that is resistant to standard treatment (prednisone and cyclophosphamide [Cytoxan]) into a new study to determine if they can be successfully treated with a blood stem cell transplantation obtained from an appropriate donor. Donors will be human leukocyte antigen (HLA)-matched healthy brothers or sisters. For patients without sibling HLA-matches, a search for donors will be initiated through the US and International Donor Registries. Eligible patients must be at least 18 years old and have SLE with progressive kidney, lung, heart, or central nervous system disease that has not responded to standard therapy.

Patients will be treated for two weeks to prepare them for the infusion of blood stem cells that are obtained from their HLA-matched donor. Patients will initially be treated with immunosuppressive drugs, which will be gradually withdrawn at approximately 6 months after transplantation. The goal of this study is to replace the abnormal immune cells of the SLE affected patient that causes the disease with normal immune cells that are generated from the transplant blood stem cells from the healthy donor.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of allogeneic blood stem cell transplantation in individuals with life-threatening SLE. A non-bone marrow ablative regimen consisting of total lymphoid irradiation (TLI) and anti-thymocyte globulin (ATG) will be used to condition the recipients for transplantation. Appropriately HLA-matched donors will undergo "mobilization" of their peripheral blood mononuclear cells using G-CSF and collection by apheresis.

The preparative regimen will consist of targeted low dose radiation of lymphoid tissue administered over a 2-week period of time. During the first week of irradiation, the patients will also receive the ATG treatment. Patients will be admitted to the in-patient service for the first 5 days of the transplant preparative regimen while receiving the ATG infusion. Patients will be discharged for the second half of the preparative regimen and followed in the out-patient clinic thereafter. Patients will start immunosuppressive treatment with cyclosporine and mycophenolate mofetil prior to the infusion of mobilized peripheral blood stem cells. The mycophenolate mofetil will be stopped at approximately 1 month post-transplantation and the cyclosporine will be tapered beginning at 2 months post-transplantation and discontinued by 6 months in the presence of stable blood chimerism and the absence of graft-versus-host disease. In the pre-transplant and post-transplant setting, patients will be evaluated by an integrated team of Rheumatology and BMT physicians. During the first 21-28 days post-transplantation, these evaluations will be performed on a daily or every other day basis. Patients will be clinically assessed and evaluated for engraftment of donor cells and disease response. Patients will then be followed as needed with maximum time between evaluations of 1 to 2 weeks in the first 100 days, and then monthly for 6 months and every 6 months to 12 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology (ACR) criteria for classification of SLE (i.e., at least 4 of the 11 criteria; see Appendix 2 of the protocol for more information)
* SLE disease activity index (SLEDAI) greater than 20 (i.e., active, multi-system SLE; see Appendix 3 of the protocol for more information)
* History of one or more of the following conditions that have not responded to conventional therapy with pulse intravenous or oral cyclophosphamide and corticosteroids:

  1. Lupus pneumonitis with a progressive decline in lung function tests and evidence of oxygen desaturation on effort in which the lung CT scans and chest X-rays show active disease without irreversible extensive scarring
  2. Diffuse alveolar hemorrhage associated with oxygen desaturation with persistent abnormalities of the lung CT scan or X-rays that have not resolved after conventional therapy
  3. Central nervous system lupus that has resulted in neurological deficits requiring hospitalization with a brain CT scan and/or brain MRI and shows evidence of lupus activity without extensive irreversible lesions
  4. Lupus nephritis with a progressive decline in the creatinine clearance that has not fallen below 25 ml/min in which a biopsy shows active disease without irreversible extensive scarring
* Refractory disease, as determined by failure of the following two conditions:

  1. Trial of corticosteroids (equivalent to prednisone 0.5 mg/kg/day for 2 months and/or at least 3 pulses of methylprednisolone 1,000 mg over 3 days) on at least one occasion within the 6 months prior to study entry
  2. Trial of cyclophosphamide of at least 500 mg/m² IV pulse at least 3 times or oral cyclophosphamide for at least 30 days
* Must have a fully HLA identical sibling or a matched unrelated donor
* Willing to use contraception throughout the study and for 12 months following treatment

Exclusion Criteria:

* Allergic to rabbit ATG
* Score of less than 60% on Karnofsky Performance Scale
* Organ dysfunction, defined as follows:

  1. Cardiac function ejection fraction less than 40% or uncontrolled malignant arrhythmias or clinical evidence of congestive heart failure (New York Class 3-4, see Appendix 4 of the protocol for more information)
  2. Pulmonary diffusion capacity (DLCO) less than 30% of predicted
  3. Liver function abnormalities with direct bilirubin levels greater than 3.0 mg/dL on two repeated tests and/or transaminases greater than 4 times the upper limit of normal
  4. Measured creatinine clearance of less than 40 ml/min (24 hour urine collection)
* Pregnant

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2004-06 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Time to achieve complete remission (participants that are off all immunosuppressive therapy without clinical or laboratory evidence of active disease) | Measured within the first year

SECONDARY OUTCOMES:
Percentage of patients with stable chimerism in all blood and immune cell lineages | Measured within the first year
Percentage of participants with acute or chronic graft-versus-host disease | Measured within the first year

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Shizuru, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No